CLINICAL TRIAL: NCT01784861
Title: A Phase I/II Study of X-82, an Oral Anti-VEGFR Tyrosine Kinase Inhibitor, With Everolimus for Patients With Pancreatic Neuroendocrine Tumors
Brief Title: VEGFR/PDGFR Dual Kinase Inhibitor X-82 and Everolimus for Treating Patients With Pancreatic Neuroendocrine Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company decision
Sponsor: Washington University School of Medicine (Other)
Collaborators: Tyrogenex (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201303150
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Adenocarcinoma; Pancreatic Neoplasms
MeSH Terms: conditions — Adenocarcinoma; Pancreatic Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase I Dose Level 0: X-82 + Everolimus (Experimental): * X-82 100 mg by mouth once daily
  * Everolimus 10mg by mouth once daily for each cycle
  * Everolimus and X-82 should be taken at the same time every day
  * 28 days =1 cycle
  Interventions: Drug: X-82; Drug: Everolimus
- Phase I Dose Level 1: X-82 + Everolimus (Experimental): * X-82 150 mg by mouth once daily
  * Everolimus 10mg by mouth once daily for each cycle
  * Everolimus and X-82 should be taken at the same time every day
  * 28 days =1 cycle
  Interventions: Drug: X-82; Drug: Everolimus
- Phase I Dose Level 2: X-82 + Everolimus (Experimental): * X-82 200 mg by mouth once daily
  * Everolimus 10mg by mouth once daily for each cycle
  * Everolimus and X-82 should be taken at the same time every day
  * 28 days =1 cycle
  Interventions: Drug: X-82; Drug: Everolimus
- Phase II: X-82 + Everolimus (Experimental): * X-82 (dose determined by Phase I portion to be 300 mg) mg by mouth once daily
  * Everolimus 10mg by mouth once daily for each cycle
  * 28 days =1 cycle
  Interventions: Drug: X-82; Drug: Everolimus
- Phase I Dose Level 3: X-82 + Everolimus (Experimental): * X-82 300 mg by mouth once daily
  * Everolimus 10mg by mouth once daily for each cycle
  * Everolimus and X-82 should be taken at the same time every day
  * 28 days =1 cycle
  Interventions: Drug: X-82; Drug: Everolimus
- Phase I Dose Level 4: X-82 + Everolimus (Experimental): * Everolimus 10mg by mouth once daily for each cycle MUST BE TAKEN FIRST
  * X-82 400 mg by mouth once daily 2 HOURS AFTER everolimus dose
  * 28 days =1 cycle
  Interventions: Drug: X-82; Drug: Everolimus

INTERVENTIONS:
Drug: X-82
  Other Names: Afinitor®; Afinitor Disperz®
Drug: Everolimus
  Other Names: Zortress®; RAD001

SUMMARY:
This study is to evaluate the combination of an investigational drug X-82 with everolimus in the treatment of pancreatic neuroendocrine tumors.

ELIGIBILITY:
Inclusion Criteria:

Phase I and PK Expansion Cohort Inclusion Criteria

* Phase I Patients: Histologic documentation of a solid malignancy and has exhausted available standard medical treatments or has no standard treatments currently available. This includes primary brain tumors.
* PK Expansion Patients: Histologic documentation of locally unresectable or metastatic renal cell carcinoma not currently amenable to surgery, radiation, or other therapy with curative intent.
* Measurable or nonmeasurable disease per RECIST 1.1 criteria.
* ECOG performance status of 0-1
* At least 18 years of age.
* Normal bone marrow and organ function as defined below:

  * Granulocytes ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥9 g/dL
  * Creatinine ≤ 1.5 x ULN
  * Bilirubin ≤ 1.5 x ULN
  * AST and ALT ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present)
  * Urine protein ≤ 1+ OR urine protein to creatinine ratio ≤ 1; if UPC ratio is > 1 on urinalysis, then 24-hour urine collection for protein must be obtained and level must be < 1,000 mg for patient enrollment.
* QTcF < 450 ms.
* Normal LVEF.
* Recovery from any major or minor surgeries.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to swallow and retain oral medication.
* Able to understand and willing to sign written informed consent document.

Phase II Inclusion Criteria

* Histologic documentation of well differentiated or moderately differentiated locally unresectable or metastatic pancreatic neuroendocrine tumor from either a primary or metastatic site with documented disease progression ≤ 12 months prior to enrollment whose disease is not currently amenable to surgery, radiation, or other modality therapy with curative intent. If different histologic classification schemes are used, equivalent histologic classifications (for example "grade 1," "low grade," or "intermediate grade") are allowed. There must be histologic documentation of a pancreatic primary site or clinical evidence of a pancreatic neuroendocrine primary tumor as determined by the treating physician. Documentation from a metastatic site is sufficient if there is clinical evidence of a pancreatic primary site. In the case of discordant pathology, patient eligibility will be determined by the PI after review of available records. Patients with neuroendocrine tumors (e.g., gastrinoma, VIPoma) in whom a pancreatic or peripancreatic primary site is strongly suspected are also eligible.
* Evidence of measurable disease per RECIST 1.1. Measurable disease is defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 2 cm with conventional techniques or as ≥ 1 cm with spiral CT scan.
* There is no limit on the number of prior chemotherapy regimens allowed. Any prior treatment (with the exception of lanreotide or octreotide) must be completed at least 4 weeks prior to initiation of treatment.
* Prior treatment with embolization or ablative therapies is allowed if measurable disease remains outside of the treated area or if there is definite progression of the treated lesions. There is no limit on the number of prior procedures.
* ECOG performance status of 0-1
* At least 18 years of age.
* Normal bone marrow and organ function as defined below:

  * Granulocytes ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥9 g/dL
  * Creatinine ≤ 1.5 x ULN
  * Bilirubin ≤ 1.5 x ULN
  * ALT and AST ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases are present)
  * Urine protein ≤ 1+ OR urine protein to creatinine ratio ≤ 1; if UPC ratio is > 1 on urinalysis, then 24-hour urine collection for protein must be obtained and level must be < 1,000 mg for patient enrollment.
* QTcF < 450 ms.
* Normal LVEF.
* Patients with fasting serum cholesterol > 300 mg/dL OR > 7.75 mmol/L AND fasting triglycerides > 2.5 x ULN should initiate lipid lowering medications.
* Recovery from any major or minor surgeries. Patient must be 4 weeks post-major surgery and 2 weeks post-minor surgery.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to swallow and retain oral medication.
* Able to understand and willing to sign written informed consent document.

Exclusion Criteria:

Phase I and PK Expansion Cohort Exclusion Criteria

* Active or severe liver disease (acute or chronic hepatitis, cirrhosis).
* Patients currently receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization).
* Receiving any other investigational agent(s) within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. A minimum of 10 days between termination of the investigational drug and administration of study drug is required.
* Any radiotherapy or immunotherapy within the last 3 weeks (limited palliative radiation is allowed ≥2 weeks). Chemotherapy regimens with delayed toxicity within the last 4 weeks (or within the last 6 weeks for prior nitrosourea or mitomycin C). Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
* Major surgery within the last 4 weeks; minor surgery within the last 2 weeks.
* Immunization with any attenuated live vaccine within 1 week prior to registration.
* Concurrent condition resulting in immune compromise, including chronic treatment with corticosteroids or other immunosuppressive agents.
* History of allergic reactions attributed to, or intolerance of, or other significant toxicity with, compounds of similar chemical or biologic composition to X-82 or everolimus.
* Patients with fasting serum cholesterol > 300 mg/dL OR > 7.75 mmol/L AND fasting triglycerides > 2.5 x ULN who would need to initiate lipid lowering medications.
* Concomitant use of drugs with a risk of causing prolonged QTc and/or Torsades de Pointes, or patients with a history of risk factors for Torsades de Pointes (e.g., familial long QT syndrome, heart failure, left ventricular hypertrophy, slow heart rate (<45 beats per minute)).
* Concomitant use of herbal medications (i.e. St. John's wort, Kava, ephedra (ma huang), ginkgo biloba) at least 7 days prior to the first dose of study drug and throughout participation in the trial.
* Concomitant use of any drug which is a moderate or strong CYP3A4 inhibitor or strong CYP3A4 inducer.
* Patients with known CNS metastases, unless metastases are treated and stable and the patients do not require systemic steroids.
* Treatment with therapeutic doses of coumarin-type anticoagulants (maximum daily dose of 1 mg allowed for port line patency permitted). Low molecular weight heparin (LMWH) will be allowed.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, inadequately controlled hypertension, uncontrolled diabetes mellitus, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or cerebrovascular accident or transient ischemic attack within 6 months of starting study drugs, or psychiatric illness/social situations that would limit compliance with study requirements.
* Presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of the study drugs.
* Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.
* Pregnant or breastfeeding.
* Known HIV-positivity on combination antiretroviral because of the potential for pharmacokinetic interactions with X-82 or everolimus. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Phase II Exclusion Criteria

* Poorly differentiated neuroendocrine carcinoma or small cell carcinoma.
* Prior treatment with everolimus, other mTOR inhibitors, or anti-VEGF drug (sunitinib, bevacizumab).
* Patients currently receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery and/or tumor embolization).
* Major surgery < 4 weeks from the start of treatment.
* Minor surgery < 2 weeks from the start of treatment. (Insertion of a vascular access device is not considered major or minor surgery.)
* Any radiotherapy or immunotherapy within the last 21 days (limited palliative radiation is allowed ≥2 weeks). Chemotherapy regimens with delayed toxicity within the last 4 weeks. Chemotherapy regimens given continuously or on a weekly basis with limited potential for delayed toxicity within the last 2 weeks.
* Immunization with any attenuated live vaccine within 1 week prior to registration.
* Concurrent condition resulting in immune compromise, including chronic treatment with corticosteroids or other immunosuppressive agents.
* Concomitant use of drugs with a risk of causing prolonged QTc and/or Torsades de Pointes, or patients with a history of risk factors for Torsades de Pointes (e.g., familial long QT syndrome, heart failure, left ventricular hypertrophy, slow heart rate (<45 beats per minute)).
* Concomitant use of herbal medications (i.e. St. John's wort, Kava, ephedra (ma huang), ginkgo biloba) at least 7 days prior to the first dose of study drug and throughout participation in the trial.
* Concomitant use of any drug which is a moderate or strong CYP3A4 inhibitor or strong CYP3A4 inducer.
* Active or severe liver disease (acute or chronic hepatitis, cirrhosis).
* Positive anti-HBV. HBV seropositive patients (HBsAg positive) are eligible if they are closely monitored for evidence of active HBV infection by HBV DNA testing, and they must agree to receive suppressive therapy with lamivudine or other HBV-suppressive therapy until at least 4 weeks after the last dose of everolimus. Patients who are anti-HCV positive are eligible provided that hepatitis C viral load (hepatitis C RNA) is undetectable.
* Clinical evidence of brain metastases or carcinomatous meningitis.
* History of GI perforation within 12 months prior to registration or presence of active gastrointestinal (GI) disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of the study drugs.
* History of clinically significant bleeding episodes.
* Current NYHA class II, III, or IV congestive heart failure (see Appendix C) or symptomatic heart failure within 60 days prior to the start of study drugs.
* Symptomatic arterial peripheral vascular disease.
* History of aortic aneurysm, aortic dissection, angina, myocardial infarction, stroke, transient ischemic attack, or other arterial thrombotic events within 6 months of registration. Patients on therapeutic non-coumarin anticoagulation are eligible provided that they are on a stable dose of anticoagulants.
* Uncontrolled diabetes mellitus or inadequately controlled hypertension.
* Receiving any other investigational agent(s) within 21 days or 5 half-lives (whichever is shorter) prior to the first dose of study drug. A minimum of 10 days between termination of the investigational drug and administration of study drug is required.
* History of allergic reactions or intolerance of, or other significant toxicity with, attributed to compounds of similar chemical or biologic composition to X-82 or everolimus.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
* Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol
* Pregnant or breastfeeding.
* Known HIV-positivity on combination antiretroviral because of the potential for pharmacokinetic interactions with X-82 or everolimus. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05-03 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Tan, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Washington University School of Medicine, St Louis, Missouri
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pedersen KS, Grierson PM, Picus J, Lockhart AC, Roth BJ, Liu J, Morton A, Chan E, Huffman J, Liang C, Wang-Gillam A, Tan B. Vorolanib (X-82), an oral anti-VEGFR/PDGFR/CSF1R tyrosine kinase inhibitor, with everolimus in solid tumors: results of a phase I study. Invest New Drugs. 2021 Oct;39(5):1298-1305. doi: 10.1007/s10637-021-01093-7. Epub 2021 Mar 18. PMID 33738668
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level 4: X-82 + Everolimus: * Everolimus 10mg by mouth once daily for each cycle MUST BE TAKEN FIRST
  * X-82 400 mg by mouth once daily 2 HOURS AFTER everolimus dose
  * 28 days =1 cycle
  X-82
  Everolimus
Period: Overall Study
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Started | 3 | 3 | 4 | 8 | 3 | 2
Completed | 3 | 3 | 3 | 3 | 2 | 1
Not Completed | 0 | 0 | 1 | 5 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus | Total
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 3 | 2 | 23
Age, Continuous [Median (Full Range); unit: years] | 71 [49 to 72] | 61 [48 to 62] | 53 [50 to 80] | 53 [36 to 72] | 59 [55 to 73] | 64.5 [63 to 66] | 59 [36 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 2 | 2 | 0 | 11
  Male | 2 | 0 | 1 | 6 | 1 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4 | 8 | 2 | 1 | 19
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 0 | 1 | 0 | 6
  White | 1 | 1 | 3 | 8 | 1 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 8 | 3 | 2 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities - Phase I
Description: Tolerability of X-82 in combination with everolimus will be determined by NCI Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
Time Frame: Completion of 1st cycle for all patients in Phase I portion of study (completed in approximately 20 months)
Population: -1 participant in Phase I Dose Level 2 was not evaluable for this outcome measure because they received less than one cycle of treatment. 1 participant in Phase I Dose Level 3 was not evaluable for this outcome measure because they received less than one cycle of treatment. 1 participant in Phase I Dose Level 3 was not evaluable for this outcome measure because they didn't receive any treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 0
Participants | 0 | 0 | 0 | 1 | 0 |

2. Primary Outcome: Overall Toxicities - Phase I
Description: -Toxicities will be graded by the NCI Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
Time Frame: 30 days after completion of treatment (estimated to be 13 months)
Population: Phase II is zero analyzed because this outcome measure is for Phase I participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 3 | 3 | 4 | 8 | 3 | 0
Participants
  Anemia | 0 | 1 | 0 | 1 | 0 |
  Hearing impaired | 1 | 0 | 0 | 0 | 0 |
  Peripheral vision/depth perception impairment | 0 | 1 | 0 | 0 | 0 |
  Abdominal distension | 0 | 1 | 0 | 0 | 0 |
  Abdominal pain | 1 | 0 | 1 | 5 | 2 |
  Colonic fistula | 0 | 0 | 0 | 1 | 0 |
  Constipation | 0 | 1 | 1 | 1 | 0 |
  Diarrhea | 2 | 2 | 2 | 3 | 2 |
  Dry mouth | 0 | 0 | 0 | 2 | 0 |
  Dyspepsia | 0 | 1 | 0 | 0 | 0 |
  Flatulence | 0 | 0 | 1 | 1 | 0 |
  Hemorrhoids | 0 | 0 | 0 | 1 | 0 |
  Intra-abdominal hemorrhage | 0 | 1 | 0 | 0 | 1 |
  Loss of taste | 0 | 0 | 0 | 1 | 0 |
  Mucositis oral | 2 | 2 | 2 | 4 | 2 |
  Nausea | 1 | 1 | 1 | 3 | 1 |
  Rectal fissure | 0 | 0 | 0 | 1 | 0 |
  Stomach pain | 0 | 0 | 1 | 0 | 0 |
  Taste changes | 0 | 0 | 1 | 0 | 0 |
  Vomiting | 1 | 1 | 1 | 2 | 1 |
  Chills | 0 | 1 | 1 | 3 | 0 |
  Edema face | 0 | 0 | 0 | 4 | 0 |
  Edema limbs | 0 | 1 | 2 | 3 | 1 |
  Fatigue | 1 | 2 | 3 | 5 | 2 |
  Fever | 0 | 1 | 0 | 2 | 0 |
  Pain | 0 | 0 | 2 | 0 | 1 |
  Cold sores | 0 | 0 | 1 | 0 | 0 |
  Elevated lactate dehydrogenase total | 0 | 0 | 0 | 0 | 1 |
  Oral thrush | 0 | 2 | 0 | 0 | 0 |
  Peritoneal infection | 0 | 1 | 0 | 0 | 0 |
  Sinusitis | 0 | 1 | 0 | 2 | 0 |
  Upper respiratory infection | 1 | 0 | 0 | 0 | 0 |
  Urinary tract infection | 1 | 0 | 0 | 0 | 0 |
  Bruising | 0 | 0 | 0 | 2 | 0 |
  Slow wound healing | 0 | 0 | 0 | 1 | 0 |
  Alkaline phosphatase increased | 0 | 0 | 0 | 1 | 0 |
  Blood bilirubin increased | 0 | 0 | 0 | 1 | 0 |
  Creatinine increased | 0 | 0 | 0 | 1 | 1 |
  Neutrophil count decreased | 0 | 0 | 2 | 3 | 0 |
  Platelet count decreased | 0 | 0 | 0 | 4 | 0 |
  Weight loss | 1 | 0 | 1 | 1 | 0 |
  Anorexia | 1 | 1 | 3 | 3 | 3 |
  Dehydration | 1 | 0 | 0 | 0 | 2 |
  Hypernatremia | 0 | 0 | 0 | 0 | 1 |
  Hypertriglyceridemia | 0 | 0 | 0 | 2 | 1 |
  Hypophosphatemia | 0 | 0 | 0 | 1 | 0 |
  Arthralgia | 0 | 0 | 1 | 0 | 1 |
  Back pain | 0 | 1 | 1 | 2 | 0 |
  Flank pain | 0 | 1 | 1 | 1 | 0 |
  Myalgia | 0 | 0 | 0 | 1 | 0 |
  Pain to extremity | 0 | 0 | 0 | 2 | 0 |
  Aphasia | 1 | 0 | 0 | 0 | 0 |
  Dizziness | 1 | 1 | 0 | 2 | 1 |
  Dysgeusia | 0 | 0 | 0 | 2 | 1 |
  Headache | 1 | 0 | 0 | 3 | 1 |
  Tremor | 0 | 0 | 1 | 0 | 0 |
  Trigeminal nerve disorder | 0 | 0 | 1 | 0 | 0 |
  Anxiety | 0 | 0 | 1 | 0 | 0 |
  Confusion | 0 | 1 | 0 | 1 | 0 |
  Depression | 0 | 0 | 1 | 1 | 0 |
  Insomnia | 1 | 0 | 0 | 3 | 1 |
  Libido decreased | 0 | 0 | 0 | 1 | 0 |
  Mood swings | 0 | 0 | 0 | 1 | 0 |
  Hematuria | 0 | 0 | 1 | 0 | 0 |
  Urinary frequency | 0 | 0 | 0 | 2 | 0 |
  Testicular pain | 0 | 0 | 0 | 1 | 0 |
  Cough | 0 | 0 | 2 | 2 | 1 |
  Dyspnea | 1 | 1 | 1 | 1 | 1 |
  Epistaxis | 0 | 0 | 1 | 3 | 0 |
  Hiccups | 1 | 0 | 0 | 0 | 0 |
  Hypoxia | 0 | 1 | 0 | 0 | 0 |
  Nasal congestion | 0 | 0 | 0 | 1 | 0 |
  Sore throat | 0 | 0 | 1 | 0 | 0 |
  Alopecia | 0 | 0 | 1 | 0 | 0 |
  Hair color changes | 0 | 0 | 1 | 0 | 0 |
  Pruritis | 0 | 0 | 0 | 2 | 0 |
  Rash acneiform | 0 | 0 | 0 | 1 | 1 |
  Rash maculo-papular | 0 | 1 | 2 | 2 | 1 |
  Skin hypopigmentation | 0 | 1 | 1 | 0 | 0 |
  Skin thinning | 0 | 0 | 0 | 1 | 0 |
  Hot flashes | 0 | 0 | 0 | 0 | 1 |
  Hypertension | 0 | 0 | 1 | 1 | 0 |
  Dysphagia | 0 | 0 | 0 | 0 | 1 |
  Hypovolemia | 0 | 1 | 0 | 0 | 0 |
  Intraperitoneal bleeding | 0 | 1 | 0 | 0 | 0 |
  Night sweats | 1 | 0 | 0 | 0 | 0 |
  Thromboembolic event | 0 | 1 | 0 | 1 | 0 |
  Lung infection | 0 | 0 | 0 | 0 | 1 |
  Pancreas infection | 0 | 0 | 0 | 0 | 1 |
  Sepsis | 0 | 1 | 0 | 0 | 0 |
  Diabetic ketoacidosis | 0 | 1 | 0 | 0 | 0 |
  Stroke | 1 | 0 | 0 | 0 | 0 |
  Pleural effusion | 0 | 0 | 0 | 1 | 0 |
  Mesenteric ischemia | 0 | 1 | 0 | 0 | 0 |

3. Primary Outcome: Recommended Phase II Dose of X-82
Time Frame: Completion of 1st cycle for all patients in Phase I portion of study (completed in approximately 20 months)
Population: This was the recommended Phase II dose because there were concerns about the ability to maintain the 400 mg daily dosing level for multiple cycles without significant toxicity.
Measure: Number; unit: mg
Groups:
- Phase I All Dose Levels: X-82 + Everolimus: * X-82 by mouth once daily
  * Everolimus 10mg by mouth once daily for each cycle
  * Everolimus and X-82 should be taken at the same time every day
  * 28 days =1 cycle
Arm/Group | Phase I All Dose Levels: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 21 | 0
mg | 300 |

4. Primary Outcome: Objective Response Rate (Complete Response + Partial Response) - Phase II
Description: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Through completion of treatment (estimated to be 12 months)
Population: Phase I participants are not evaluable for this outcome measure. One participant in the Phase II portion of the study was not evaluable because the treating physician removed the participant from the treatment prior to receiving the end of cycle 3 imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
Participants |  |  |  |  |  | 0

5. Secondary Outcome: Disease Stabilization Rate - Phase II
Description: * Disease stabilization rate is defined as the proportion of patients achieving a best overall response of complete response, partial response, or stable disease.
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  * Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.
Time Frame: Through completion of treatment (estimated to be 12 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
Participants |  |  |  |  |  | 1

6. Secondary Outcome: Progression Free Survival (PFS) - Phase II
Description: * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Up to 3 years
Population: Phase I participants are not evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2
days |  |  |  |  |  | 183 [174 to 192]

7. Secondary Outcome: Overall Survival - Phase II
Description: Start of the treatment until death.
Time Frame: Up to 3 years
Population: Phase I participants are not evaluable for this outcome measure.
Measure: Median (Full Range); unit: days
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2
days |  |  |  |  |  | 115 [94 to 136]

8. Secondary Outcome: Number of Participants With Toxicity - Phase II
Description: Toxicity will be graded by NCI Common Terminology Criteria for Adverse Events (CTCAE version 4.0)
Time Frame: Through 30 days after completion of treatment (estimated to be 13 months)
Population: Phase I participants are not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 2
Participants
  Diarrhea |  |  |  |  |  | 2
  Mucositis oral |  |  |  |  |  | 1
  Nausea |  |  |  |  |  | 1
  Vomiting |  |  |  |  |  | 1
  Chest pain |  |  |  |  |  | 1
  Edema limbs |  |  |  |  |  | 1
  Hematoma |  |  |  |  |  | 1
  Mouth sores |  |  |  |  |  | 1
  Creatinine increased |  |  |  |  |  | 1
  Platelet count decreased |  |  |  |  |  | 1
  Hip pain |  |  |  |  |  | 1
  Leg cramps |  |  |  |  |  | 1
  Dizziness |  |  |  |  |  | 1
  Headache |  |  |  |  |  | 1
  Allergic rhinitis |  |  |  |  |  | 1
  Rash acneiform |  |  |  |  |  | 1
  Rash maculo-papular |  |  |  |  |  | 1
  Hypertension |  |  |  |  |  | 1

ADVERSE EVENTS:
Time Frame: Adverse events were followed from start of treatment through 30 days following end of treatment. All-cause mortality was followed from start of treatment through completion of follow-up.
Arm/Group | Phase I Dose Level 0: X-82 + Everolimus | Phase I Dose Level 1: X-82 + Everolimus | Phase I Dose Level 2: X-82 + Everolimus | Phase I Dose Level 3: X-82 + Everolimus | Phase I Dose Level 4: X-82 + Everolimus | Phase II: X-82 + Everolimus
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 5/8 | 2/3 | 2/2
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 0/4 | 2/8 | 2/3 | 2/2
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 8/8 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0: X-82 + Everolimus (N=3) | Phase I Dose Level 1: X-82 + Everolimus (N=3) | Phase I Dose Level 2: X-82 + Everolimus (N=4) | Phase I Dose Level 3: X-82 + Everolimus (N=8) | Phase I Dose Level 4: X-82 + Everolimus (N=3) | Phase II: X-82 + Everolimus (N=2)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oral thrush (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Pancreas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Peritoneal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypovolemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Intraperitoneal bleeding (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mesenteric ischemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 0: X-82 + Everolimus (N=3) | Phase I Dose Level 1: X-82 + Everolimus (N=3) | Phase I Dose Level 2: X-82 + Everolimus (N=4) | Phase I Dose Level 3: X-82 + Everolimus (N=8) | Phase I Dose Level 4: X-82 + Everolimus (N=3) | Phase II: X-82 + Everolimus (N=2)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral vision/depth perception impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 4 | 1 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Loss of taste (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 2 | 4 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 1 | 1
Rectal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Taste changes (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 1 | 1
Chills (General disorders) | 0 | 1 | 1 | 3 | 0 | 0
Edema face (General disorders) | 0 | 0 | 0 | 4 | 0 | 0
Edema limbs (General disorders) | 0 | 1 | 2 | 3 | 1 | 1
Fatigue (General disorders) | 1 | 2 | 3 | 5 | 2 | 0
Fever (General disorders) | 0 | 1 | 0 | 2 | 0 | 0
Pain (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Cold sores (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Elevated lactate dehydrogenase total (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Mouth sores (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Slow wound healing (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 3 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 4 | 0 | 1
Weight loss (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 3 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Hip pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain to extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 2 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 3 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 3 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hair color changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 2 | 1 | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Skin thinning (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1
Night sweats (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT01784861/Prot_SAP_000.pdf